CLINICAL TRIAL: NCT04141631
Title: Patient Blood Management in Cardiac Surgery by Erythropoietin, Ferric Carboxymaltose and Metabolic Adjustment (ScvO2): A Randomized Controlled Study
Brief Title: Transfusion Savings in Heart Surgery: Impact of Individual Strategy by Erythropoietin and Metabolic Adjustment (ScvO2)
Acronym: BLOOCOST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL19_0042
Record Dates: First submitted 2019-10-04; First posted 2019-10-28 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-09

CONDITIONS: Cardiac Surgery; Transfusion; Perioperative Anemia
Keywords: Perioperative Erythropoietin; Perioperative Iron; ScVO2; Patient blood Management; Blood Transfusion
MeSH Terms: interventions — ferric carboxymaltose; Fosfomycin; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STOP Group (Experimental): EPO (600UI/Kg, sub-cutaneous) and Ferric Carboxymaltose (FCM) (20 mg/kg in 250 mL of saline solution 0.9% over 15 min) will be administered if
  * Hb < 13g/dL the day before surgery
  * Hb ≥ 7g/dL AND ScvO2 > 65% in postoperative ICU stay
  Postoperative Transfusion will be guided by ScvO2 values :
  if Hb ≤ 8 g/dL AND ScvO2 ≤ 65% or if Hb < 7g/dL independently of ScVO2 value
  Interventions: Drug: EPO (600UI/Kg, sub-cutaneous) and Ferric Carboxymaltose (FCM) (20 mg/kg in 250 mL of saline solution 0.9% over 15 min)
- Control Group (No Intervention): Only postoperative anemia will be managed:
  * RBC transfusion will be performed if Hb ≤ 8 g/dL (2017 EACTS/EACTA guidelines)
  * Iron sucrose administration if Hb > 8g/dL : 2 injections of 200 mg according to Height (+/- 70 Kg) in 250 mL of saline solution 0.9% over 1h30 into 48 h intervals without exceeding a total dose of 15mg/kg.

INTERVENTIONS:
Drug: EPO (600UI/Kg, sub-cutaneous) and Ferric Carboxymaltose (FCM) (20 mg/kg in 250 mL of saline solution 0.9% over 15 min) — EPO (600UI/Kg, sub-cutaneous) and Ferric Carboxymaltose (FCM) (20 mg/kg in 250 mL of saline solution 0.9% over 15 min) will be administered if
  * Hb < 13g/dL the day before surgery
  * Hb ≥ 7g/dL AND ScvO2 > 65% in postoperative ICU stay
  Postoperative Transfusion will be guided by ScvO2 values :
  if Hb ≤ 8 g/dL AND ScvO2 ≤ 65% or if Hb < 7g/dL independently of ScVO2 value
  Arms: STOP Group

SUMMARY:
Preoperative anemia, bleeding and transfusions have been recognized as a "Deadly triad" in cardiac surgery associated with an increased morbidity,mortality, and costs related. Thus strategies to reduce unnecessary RBC transfusions and to optimize preoperative anemia must be developed .The study evaluate an individual blood conservation strategy based on patient blood management bundles in cardiac surgery patients: optimisation perioperative hemoglobin level by erythropoietin and ferric carboxymaltose (Ferinject) associated with the use of ScV02 to guide perioperative erythrocyte transfusion.

DETAILED DESCRIPTION:
Preoperative anemia is the most common haematological abnormalities in cardiac surgery affecting 20 to 40% of patients and is becoming increasingly prevalent due to an ageing population with more chronic diseases.Preoperative anemia is independently associated with increased risk of adverse outcome following cardiac surgery but also implies blood transfusions which, associated with anemia, increase significantly perioperative cardiac morbidity and mortality. Therefore, strategies of blood conservation to optimize anemia and to minimize transfusion have been developped in the concept of the Blood Patient Management (BPM). To correct anemia, intravenous iron has been shown to be an effective treatment with increase hemoglobin (Hb) level in the perioperative period. It is now established that intravenous iron, as ferric carboxymaltose (Ferinject) is better tolerated compared to oral supplementation with better stimulation of erythropoiesis and,consequently, higher Hb levels. Based on promising results in the orthopedic surgery patients, the use of recombinant human erythropoietin (EPO) has also been proposed in cardiac surgery. Secondly, because even one red blood cells products (RBC) compromises postoperative outcome, guidelines suggest to adopt restrictive threshold of Hb levels to decide RBC transfusion. However, beyond the fact that RBC transfusion correct Hb level, the final goal of blood transfusion is to improve oxygen delivery to hypoxemic tissue. In this respect, the relevance of the use of a Hb threshold to guide transfusion have been questioned. Venous oxygen saturation (SvO2) and ScvO2 (central oxygen venous saturation), global parameters of tissue oxygenation, in stable hemodynamic and respiratory conditions, may be an relevant marker of anemia tolerance. Recently, the investigators demonstrated the lack of benefit in terms of ScvO2 increase during erythrocyte transfusion if ScvO2 was > 65%.

In order to reduce exposure to transfusion, the management of anemia with EPO and perioperative intravenous FCM associated with the use of ScvO2 could be interesting to both improve Hb levels and reduce RBC transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled Cardiac surgery for more than 24 hours
* High risk of perioperative transfusion defined by a TRUST Score ≥ 3
* Veno-Venous catheter in Superior vena cava territory
* Patient Affiliate or beneficiary of social security
* Collection on free, informed and written consent

Exclusion Criteria:

* EPO and FCM contraindication
* Patients already treated by EPO at the time of inclusion
* Non controlled Infectious endocarditis defined by ESC guidelines 2015
* Patients including in an other research
* Patients whose physical and/or psychological health is severely impaired and who, according to the investigator, may affect the participant's compliance with the study.
* Patients deprived from his rights (guardianship or tutelage measure)
* Patients who refuses to sign the consent
* pregnant or lactating woman

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Transfusion incidence at hospital discharge | up to Day 28
  Number of patients transfused of blood units

SECONDARY OUTCOMES:
ICU transfusion incidence | at ICU discharge or up to Day 28
  Number of blood units transfused during ICU stay
total of blood units transfused | up to day 28
  number of blood units administered per patient
Hemoglobin level at surgery discharge and Hemoglobin level at 1 month after discharge from hospital | at surgery discharge (or at Day 28) and at 1 month after discharge from hospital
  the last hemoglobin value at surgery discharge and the hemoglobin value at 1 month after discharge from hospital
The total duration of mechanical ventilation | at ICU discharge or up to Day 28
  The total duration of mechanical ventilation in ICU
length of stay in ICU | up to day 28
  numbers of days in ICU
Length of hospital stay | at day 28
  Length of stay during hospitalization (Between 1 and 28 day)
Incidence of Mortality | at day 28
  Incidence of 28-day mortality
Incidence of postoperative events in ICU | at day 28
  AKI (KDIGO criteria), Cardiac dysfunction (acute heart failure requiring inotrope or extracorporeal life support (ECLS), arrythmia), vascular dysfunction (norepinephrine support without sepsis), respiratory dysfunction (non invasive ventilation devices, secondary intubation,mechanical ventilation more than 12 hours), septic complications (sepsis/septic shock)

CONTACTS AND LOCATIONS:
Locations (1):
- DEpartement d'anesthésie et réanimation D - Arnaud de Villeneuve, Montpellier, France

REFERENCES:
- [Background] Ranucci M, Baryshnikova E, Castelvecchio S, Pelissero G; Surgical and Clinical Outcome Research (SCORE) Group. Major bleeding, transfusions, and anemia: the deadly triad of cardiac surgery. Ann Thorac Surg. 2013 Aug;96(2):478-85. doi: 10.1016/j.athoracsur.2013.03.015. Epub 2013 May 11. PMID 23673069
- [Background] Plicht B, Lind A, Erbel R. [Infective endocarditis : New ESC guidelines 2015]. Internist (Berl). 2016 Jul;57(7):675-90. doi: 10.1007/s00108-016-0086-y. German. PMID 27307162
- [Background] Alghamdi AA, Davis A, Brister S, Corey P, Logan A. Development and validation of Transfusion Risk Understanding Scoring Tool (TRUST) to stratify cardiac surgery patients according to their blood transfusion needs. Transfusion. 2006 Jul;46(7):1120-9. doi: 10.1111/j.1537-2995.2006.00860.x. PMID 16836558
- [Background] Task Force on Patient Blood Management for Adult Cardiac Surgery of the European Association for Cardio-Thoracic Surgery (EACTS) and the European Association of Cardiothoracic Anaesthesiology (EACTA); Boer C, Meesters MI, Milojevic M, Benedetto U, Bolliger D, von Heymann C, Jeppsson A, Koster A, Osnabrugge RL, Ranucci M, Ravn HB, Vonk ABA, Wahba A, Pagano D. 2017 EACTS/EACTA Guidelines on patient blood management for adult cardiac surgery. J Cardiothorac Vasc Anesth. 2018 Feb;32(1):88-120. doi: 10.1053/j.jvca.2017.06.026. Epub 2017 Sep 30. No abstract available. PMID 29029990
- [Derived] Saour M, Blin C, Zeroual N, Mourad M, Amico M, Gaudard P, Picot MC, Colson PH. Impact of a bundle of care (intravenous iron, erythropoietin and transfusion metabolic adjustment) on post-operative transfusion incidence in cardiac surgery: a single-centre, randomised, open-label, parallel-group controlled pilot trial. Lancet Reg Health Eur. 2024 Jun 24;43:100966. doi: 10.1016/j.lanepe.2024.100966. eCollection 2024 Aug. PMID 39022429